CLINICAL TRIAL: NCT02756689
Title: Outpatient Foley for Starting Induction of Labor at Term
Acronym: OFFSITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Spencer G. Kuper, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F151022005
Record Dates: First submitted 2016-04-11; First posted 2016-04-29 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Pregnancy
Keywords: Mechanical cervical ripening; Transcervical catheter; Foley catheter for labor induction; Cervical ripening; Induction of labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inpatient cervical Ripening (Active Comparator): Subjects in this arm will be seen in the outpatient setting, and if they qualify and are randomized to the inpatient (control) group, they will be admitted to labor and delivery the next day for cervical ripening with a transcervical Foley catheter.
  Interventions: Other: Inpatient cervical ripening
- Outpatient cervical Ripening (Active Comparator): Subjects in this arm will undergo cervical ripening with a transcervical Foley catheter in the outpatient setting (treatment arm). The transcervical catheter will be placed in the office after confirmation of fetal well-being. They will then return the next morning to be admitted to labor and delivery for oxytocin administration.
  Interventions: Other: Outpatient cervical ripening

INTERVENTIONS:
Other: Inpatient cervical ripening — Subjects will undergo cervical ripening in the inpatient setting.
  Arms: Inpatient cervical Ripening
Other: Outpatient cervical ripening — Subjects will undergo cervical ripening in the outpatient setting. The patients will then be scheduled to return the next morning for induction of labor.
  Arms: Outpatient cervical Ripening

SUMMARY:
The investigators are performing a randomized controlled-trial investigating starting cervical ripening in the outpatient setting with a mechanical method, the transcervical Foley catheter. This is a pilot study to establish the efficacy of this method in decreasing time as in inpatient and evaluate patient satisfaction.

DETAILED DESCRIPTION:
Induction of labor is necessary in one-fourth of women and a large proportion requires cervical ripening. Cervical ripening is necessary to shorten the time to delivery and increases the chances of a vaginal delivery.

Outpatient cervical ripening is an attractive alternative to women and physicians because of the decreased amount of time spent in the hospital and opportunity for patients to be in the comforts of their home.

The investigators will conduct a randomized controlled trial comparing outpatient to inpatient cervical ripening using a transcervical Foley catheter. Women will be randomized to undergo inpatient or outpatient transcervical Foley catheter cervical ripening beyond their 39th week of gestation. Women and their infants will be followed until the time of their discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Multiparous
* Singleton gestation
* Gestational age between 39+0 and 42+0
* Vertex presentation
* Cervix ≤ 3 cm. If cervix is between 2 and 3 cm dilated, it must be <80% effaced
* No prior cesarean section or uterine surgery
* Resides within Jefferson County, Alabama.
* Access to a telephone
* Reliable transportation

Exclusion Criteria:

* Unsuitable for outpatient Foley placement management (IUGR, oligohydramnios, prior cesarean delivery, gestational hypertension, preeclampsia, or uncontrolled chronic hypertension, complex maternal disease, provider discretion). Any patient with pregestational or gestational diabetes on medications will be excluded.
* Latex allergy
* Contraindication to induction of labor
* Evidence of labor
* Fetal anomaly or demise
* Inability to given consent (non-English speaking, inability to read or write)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spencer G Kuper, MD, Principal Investigator — UAB, Department of Maternal-Fetal Medicine
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO Recommendations for Induction of Labour. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK131963/ PMID 23586118
- [Background] Kelly AJ, Alfirevic Z, Ghosh A. Outpatient versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2013 Nov 12;(11):CD007372. doi: 10.1002/14651858.CD007372.pub3. PMID 24222365
- [Background] Wing DA. Labor induction with misoprostol. Am J Obstet Gynecol. 1999 Aug;181(2):339-45. doi: 10.1016/s0002-9378(99)70558-2. PMID 10454679
- [Background] Alfirevic Z, Kelly AJ, Dowswell T. Intravenous oxytocin alone for cervical ripening and induction of labour. Cochrane Database Syst Rev. 2009 Oct 7;2009(4):CD003246. doi: 10.1002/14651858.CD003246.pub2. PMID 19821304
- [Background] Jozwiak M, Bloemenkamp KW, Kelly AJ, Mol BW, Irion O, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD001233. doi: 10.1002/14651858.CD001233.pub2. PMID 22419277
- [Background] Farmer KC, Schwartz WJ 3rd, Rayburn WF, Turnbull G. A cost-minimization analysis of intracervical prostaglandin E2 for cervical ripening in an outpatient versus inpatient setting. Clin Ther. 1996 Jul-Aug;18(4):747-56; discussion 702. doi: 10.1016/s0149-2918(96)80224-4. PMID 8879901
- [Background] Dowswell T, Kelly AJ, Livio S, Norman JE, Alfirevic Z. Different methods for the induction of labour in outpatient settings. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD007701. doi: 10.1002/14651858.CD007701.pub2. PMID 20687092
- [Background] O'Brien JM, Mercer BM, Cleary NT, Sibai BM. Efficacy of outpatient induction with low-dose intravaginal prostaglandin E2: a randomized, double-blind, placebo-controlled trial. Am J Obstet Gynecol. 1995 Dec;173(6):1855-9. doi: 10.1016/0002-9378(95)90440-9. PMID 8610775
- [Background] McKenna DS, Costa SW, Samuels P. Prostaglandin E2 cervical ripening without subsequent induction of labor. Obstet Gynecol. 1999 Jul;94(1):11-4. doi: 10.1016/s0029-7844(99)00244-6. PMID 10389710
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] Edwards RK, Szychowski JM, Berger JL, Petersen M, Ingersoll M, Bodea-Braescu AV, Lin MG. Foley catheter compared with the controlled-release dinoprostone insert: a randomized controlled trial. Obstet Gynecol. 2014 Jun;123(6):1280-1287. doi: 10.1097/AOG.0000000000000238. PMID 24807327
- [Background] Pettker CM, Pocock SB, Smok DP, Lee SM, Devine PC. Transcervical Foley catheter with and without oxytocin for cervical ripening: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1320-6. doi: 10.1097/AOG.0b013e31817615a0. PMID 18515515
- [Background] Sciscione AC, Bedder CL, Hoffman MK, Ruhstaller K, Shlossman PA. The timing of adverse events with Foley catheter preinduction cervical ripening; implications for outpatient use. Am J Perinatol. 2014 Oct;31(9):781-6. doi: 10.1055/s-0033-1359718. Epub 2013 Dec 17. PMID 24347259
- [Background] Henry A, Madan A, Reid R, Tracy SK, Austin K, Welsh A, Challis D. Outpatient Foley catheter versus inpatient prostaglandin E2 gel for induction of labour: a randomised trial. BMC Pregnancy Childbirth. 2013 Jan 29;13:25. doi: 10.1186/1471-2393-13-25. PMID 23356673
- [Background] McMaster K, Sanchez-Ramos L, Kaunitz AM. Evaluation of a Transcervical Foley Catheter as a Source of Infection: A Systematic Review and Meta-analysis. Obstet Gynecol. 2015 Sep;126(3):539-551. doi: 10.1097/AOG.0000000000001002. PMID 26244535
- [Result] Sciscione AC, Muench M, Pollock M, Jenkins TM, Tildon-Burton J, Colmorgen GH. Transcervical Foley catheter for preinduction cervical ripening in an outpatient versus inpatient setting. Obstet Gynecol. 2001 Nov;98(5 Pt 1):751-6. doi: 10.1016/s0029-7844(01)01579-4. PMID 11704164
- [Derived] Alfirevic Z, Gyte GM, Nogueira Pileggi V, Plachcinski R, Osoti AO, Finucane EM. Home versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007372. doi: 10.1002/14651858.CD007372.pub4. PMID 32852803
- [Derived] Kuper SG, Jauk VC, George DM, Edwards RK, Szychowski JM, Mazzoni SE, Wang MJ, Files P, Tita AT, Subramaniam A, Harper LM. Outpatient Foley Catheter for Induction of Labor in Parous Women: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jul;132(1):94-101. doi: 10.1097/AOG.0000000000002678. PMID 29889751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One additional patient was already scheduled to participate when the study met the projected number (128). The final (#129 patient) was offered participation in the study since she had already been scheduled for a study visit and possible induction of labor.
Groups:
- Inpatient Group: Subjects in this arm will be seen in the outpatient setting, and if they qualify and are randomized to the inpatient (control) group, they will be admitted to labor and delivery the next day for cervical ripening with a transcervical Foley catheter.
  Inpatient cervical ripening: Subjects will undergo cervical ripening in the inpatient setting.
- Outpatient Group (Intervention): Subjects in this arm will undergo cervical ripening with a transcervical Foley catheter in the outpatient setting (treatment arm). The transcervical catheter will be placed in the office after confirmation of fetal well-being. They will then return the next morning to be admitted to labor and delivery for oxytocin administration.
  Outpatient cervical ripening: Subjects will undergo cervical ripening in the outpatient setting. The patients will then be scheduled to return the next morning for induction of labor.
Period: Overall Study
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Started | 64 | 65
Completed | 64 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inpatient Group | Outpatient Group (Intervention) | Total
Number analyzed (Participants) | 64 | 65 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (4.2) | 26.6 (4.3) | 26.2 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 65 | 129
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity | 64 | 65 | 129
  Black | 58 | 55 | 113
  White | 5 | 8 | 13
  Hispanic | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 64 | 65 | 129

OUTCOME MEASURES:

1. Primary Outcome: Total Time From Admission to Delivery
Time Frame: From baseline to the time of delivery (baseline is from admission), up to 7 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
hours | 13.5 (7.0) | 12.4 (7.4)
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.38, t-test, 2 sided

2. Secondary Outcome: Total Hospital Duration
Time Frame: From admission time to the hospital until discharge from the hospital, up to 7 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
days | 2.7 (0.6) | 2.6 (0.5)
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.29, t-test, 2 sided

3. Secondary Outcome: Number of Participants Using Acetaminophen
Time Frame: From placement of Foley bulb to 24 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Participants | 6 | 13
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.09, Chi-squared; Risk Ratio (RR) = 2.1, 95% CI 2-sided [0.8 to 5.3]

4. Secondary Outcome: Number of Participants Calling the Obstetrical Triage Unit
Time Frame: From placement of Foley bulb to 24 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Participants | 0 | 4
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.12, Chi-squared

5. Secondary Outcome: Number of Participants Admitted Prior to the Scheduled Induction of Labor Time
Time Frame: From placement of Foley bulb to 24 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Participants | 3 | 10
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.06, Chi-squared; Risk Ratio (RR) = 3.3, 95% CI 2-sided [0.9 to 11.4]

6. Secondary Outcome: Number of Participants With Spontaneous Rupture of Membranes Between Foley Bulb Placement and Admission
Time Frame: From placement of Foley bulb to 24 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Participants | 5 | 4
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.74, Chi-squared; Risk Ratio (RR) = 0.8, 95% CI 2-sided [0.2 to 2.8]

7. Secondary Outcome: Nonreassuring Fetal Heart Tracings 30-minutes After Foley Bulb Placement.
Time Frame: From placement until 30 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Participants | 0 | 0
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 1, Chi-squared

8. Secondary Outcome: Total Duration of Time of Neuraxial Anesthesia Use
Time Frame: Assessed from baseline to delivery, up to 3 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
hours | 8.7 (6.3) | 8.4 (6.9)
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.82, t-test, 2 sided

9. Secondary Outcome: Total Duration of Time From Rupture of Membranes Until Delivery
Time Frame: Assessed from baseline to delivery, up to 3 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
hours | 6.2 (4.4) | 5.5 (4.4)
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.38, t-test, 2 sided

10. Secondary Outcome: Maximum Oxytocin Rate
Time Frame: Assessed from baseline to delivery, up to 3 days
Measure: Mean (Standard Deviation); unit: milliunits/min
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
milliunits/min | 16.4 (9) | 17.8 (9.6)
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.42, t-test, 2 sided

11. Secondary Outcome: Highest Maternal Intrapartum Temperature
Time Frame: Assessed from baseline to delivery, up to 3 days
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Celsius | 36.8 (0.4) | 36.7 (0.5)
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.06, t-test, 2 sided

12. Secondary Outcome: Number of Participants With Chorioamnionitis
Time Frame: Assessed from baseline to delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Participants | 3 | 3
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p > 0.99, Chi-squared; Risk Ratio (RR) = 1, 95% CI 2-sided [0.2 to 4.7]

13. Secondary Outcome: Number of Participants With Meconium-stained Fluid
Time Frame: Assessed from baseline to delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Participants | 11 | 8
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.43, Chi-squared; Risk Ratio (RR) = 0.7, 95% CI 2-sided [0.3 to 1.7]

14. Secondary Outcome: Number of Participants With Neonates With Shoulder Dystocia
Time Frame: Assessed at delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Participants | 7 | 2
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.09, Chi-squared; Risk Ratio (RR) = 0.3, 95% CI 2-sided [0.1 to 1.3]

15. Secondary Outcome: Number of Participants Who Had a Cesarean Delivery
Time Frame: Assessed from baseline to delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Participants | 3 | 2
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.68, Chi-squared; Risk Ratio (RR) = 0.7, 95% CI 2-sided [0.1 to 3.8]

16. Secondary Outcome: Number of Participants With an Operative Vaginal Delivery
Time Frame: Assessed at delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Participants | 6 | 5
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.73, Chi-squared; Risk Ratio (RR) = 0.8, 95% CI 2-sided [0.3 to 2.6]

17. Secondary Outcome: Postpartum Hemorrhage
Time Frame: Assessed at delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Participants | 1 | 0
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.5, Chi-squared

18. Secondary Outcome: Number of Participants With Endometritis
Time Frame: Assessed from delivery until 30 days post-discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Participants | 1 | 1
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p > 0.99, Chi-squared; Risk Ratio (RR) = 1, 95% CI 2-sided [0.1 to 15.4]

19. Secondary Outcome: Number of Participants With Readmission Within 30 Days
Time Frame: Assessed from time of discharge until 30 days post-discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Participants | 0 | 1
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p > 0.99, Chi-squared

20. Secondary Outcome: Number of Neonates With a 5-minute Apgar Score Less Than 7
Description: Apgar scores are assigned to all births. These are universally performed and assigned in the United States. The scoring system is between 0-10. 0 is the minimum score and 10 is the maximum. Lower scores are worse than higher scores.
Time Frame: Assessed at time of delivery up to 5-minutes post-delivery.
Measure: Number; unit: Neonates
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
Neonates | 1 | 0
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.5, Chi-squared

21. Secondary Outcome: Number of Neonates With Umbilical Artery Cord pH < 7.1
Time Frame: Assessed at time of delivery up to 5-minutes post-delivery.
Measure: Number; unit: neonates
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
neonates | 4 | 1
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.37, Chi-squared; Risk Ratio (RR) = 0.3, 95% CI 2-sided [0.03 to 2.3]

22. Secondary Outcome: Number of Neonates With an Umbilical Cord Artery Base Deficit Less Than Negative 12
Description: Base deficit is a lab value.
Time Frame: Assessed at time of delivery up to 5-minutes post-delivery.
Measure: Number; unit: neonates
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
neonates | 1 | 0
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p > 0.99, Chi-squared

23. Secondary Outcome: Number of Neonates With Birth Injuries
Description: Cephalohematomas, subgaleal hematomas, fracture of the clavicle, and scalp lacerations
Time Frame: Assessed at time of delivery up to time of neonatal discharge, up to 30 days.
Measure: Number; unit: neonates
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
neonates | 2 | 1
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p = 0.62, Chi-squared; Risk Ratio (RR) = 0.5, 95% CI 2-sided [0.05 to 5.3]

24. Secondary Outcome: Number of Neonates Admitted to the Neonatal Intensive Care Unit Admissions
Description: The rates of neonatal intensive care unit admissions will be calculated.
Time Frame: Assessed at time of delivery up to time of neonatal discharge, up to 30-days
Measure: Number; unit: neonates
Arm/Group | Inpatient Group | Outpatient Group (Intervention)
Number analyzed (Participants) | 64 | 65
neonates | 5 | 5
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group (Intervention); Test type: Superiority; p > 0.99, Chi-squared; Risk Ratio (RR) = 1, 95% CI 2-sided [0.3 to 3.2]

25. Secondary Outcome: Patient Satisfaction Six Simple Questions, Q1
Description: Assessed through validated survey, Six Simple Questions. Adapted from Harvey S, Rach D, et al. Evaluation of satisfaction with midwifery care. 2002 Dec; 18(4):260-7.
  1=strongly agree, 4 = neutral, 7=strongly agree.
  Title: Six simple questions Definition: A survey to assess patient satisfaction during their cervical ripening and induction.
  Ranges: 1-7 Best score: 7 Worst score: 1
Time Frame: At discharge.
Population: Title: Six simple questions Definition: A survey to assess patient satisfaction during their cervical ripening and induction.
  Ranges: 1-7 Best score: 7 Worst score: 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Outpatient Group: Six Simple Questions: I had appropriate consideration for my time.
- Inpatient Group: Six Simple Questions: I had appropriate and adequate control over my care.
Arm/Group | Outpatient Group | Inpatient Group
Number analyzed (Participants) | 65 | 64
units on a scale | 7 [7 to 7] | 7 [6 to 7]
Statistical Analysis 1: Comparison: Outpatient Group vs Inpatient Group; Test type: Superiority; p = 0.234, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: Patient Satisfaction (Six Simple Questions, Question 2)
Description: Assessed through validated survey (Six simple questions, Q-2). Question 2: The person(s) responsible for my care are/were caring and compassionate. Scale 1-7. 1=strongly agree, 4 = neutral, 7=strongly agree.
  Title: Six simple questions Definition: A survey to assess patient satisfaction during their cervical ripening and induction.
  Ranges: 1-7 Best score: 7 Worst score: 1
Time Frame: At discharge
Population: as for outcome 25
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group: Six Simple Questions Survey: The persons responsible for my care are/were caring and compassionate.
- Outpatient Group: Six Simple Questions: The persons responsible for my care are/were caring and compassionate.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 7 [7 to 7] | 7 [7 to 7]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Patient Satisfaction (Six Simple Questions, Question 3)
Description: Assessed through validated survey, Six Simple Questions. Adapted from Harvey S, Rach D, et al. Evaluation of satisfaction with midwifery care. 2002 Dec; 18(4):260-7.
  Question 3: Problems that have arisen up to now have not been dealt with effectively. Scale 1-7. 1=strongly agree, 4 = neutral, 7=strongly agree.
  Title: Six simple questions Definition: A survey to assess patient satisfaction during their cervical ripening and induction.
  Ranges: 1-7 Best score: 7 Worst score: 1
Time Frame: At discharge
Population: as for outcome 25
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Six Simple Questions Survey: Problems that have arisen up to now have not been dealt with effectively.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 1 [1 to 1.5] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.77, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: Patient Satisfaction (Six Simple Questions, Question 4)
Description: Assessed through validated survey, Six Simple Questions. Adapted from Harvey S, Rach D, et al. Evaluation of satisfaction with midwifery care. 2002 Dec; 18(4):260-7.
  Question 4: My needs have been addressed with appropriate consideration for my time. Scale 1-7. 1=strongly agree, 4 = neutral, 7=strongly agree.
  Title: Six simple questions Definition: A survey to assess patient satisfaction during their cervical ripening and induction.
  Ranges: 1-7 Best score: 7 Worst score: 1
Time Frame: At discharge
Population: as for outcome 25
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Six Simple Questions Survey: My needs have been addressed with appropriate consideration for my time.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 7 [7 to 7] | 7 [7 to 7]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney)

29. Secondary Outcome: Patient Satisfaction (Six Simple Questions, Question 5)
Description: Assessed through validated survey, Six Simple Questions. Adapted from Harvey S, Rach D, et al. Evaluation of satisfaction with midwifery care. 2002 Dec; 18(4):260-7.
  Question 5: The overall organization of my ca re has not been appropiate. Scale 1-7. 1=strongly agree, 4 = neutral, 7=strongly agree.
  Title: Six simple questions Definition: A survey to assess patient satisfaction during their cervical ripening and induction.
  Ranges: 1-7 Best score: 7 Worst score: 1
Time Frame: At discharge
Population: as for outcome 25
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Six Simple Questions Survey: The overall organization of my care has not been appropriate.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 1 [1 to 1] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.75, Wilcoxon (Mann-Whitney)

30. Secondary Outcome: Patient Satisfaction (Six Simple Questions, Question 6)
Description: Assessed through validated survey, Six Simple Questions. Adapted from Harvey S, Rach D, et al. Evaluation of satisfaction with midwifery care. 2002 Dec; 18(4):260-7.
  Question 6: I would choose the same type of care for my next pregnancy. Scale 1-7. 1=strongly agree, 4 = neutral, 7=strongly agree.
  Title: Six simple questions Definition: A survey to assess patient satisfaction during their cervical ripening and induction.
  Ranges: 1-7 Best score: 7 Worst score: 1
Time Frame: At discharge
Population: as for outcome 25
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Six Simple Questions Survey: I would choose the same type of care for my next pregnancy.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 7 [6 to 7] | 7 [7 to 7]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.75, Wilcoxon (Mann-Whitney)

31. Secondary Outcome: Patient Satisfaction (Lady-X Survey, Question 1)
Description: Assessed through a validated survey, Lady-X. Adapted from Gartner FR, de Bekker-Grob EW et al. Calculating preference weights for the labor and delivery index: A discrete choice experiment on women's birth experiences. Value Health. 2015 Sep; 856-864.
  Question 1: Presence of healthcare professionals during my birth. Scale 1-3. 1 = At all times, 2 = Most of the time, 3 = rarely
  Title: Lady-X Survey Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction.
  Ranges: 1-3 Best score: 1 Worst score: 3
Time Frame: At discharge
Population: Title: Lady-X Survey Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction.
  Ranges: 1-3 Best score: 1 Worst score: 3
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Lady-X Survey: Presence of expert healthcare professionals during my childbirth.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 1 [1 to 1] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney)

32. Secondary Outcome: Patient Satisfaction (Lady-X Survey, Question 2)
Description: Assessed through a validated survey, Lady-X Survey. Adapted from Gartner FR, de Bekker-Grob EW et al. Calculating preference weights for the labor and delivery index: A discrete choice experiment on women's birth experiences. Value Health. 2015 Sep; 856-864.
  Question 2: Information given by the healthcare professionals during childbirth. Scale 1-3. 1 = I felt very well informed by the healthcare professionals, 2 = I felt adequately informed by the healthcare professionals, 3 = I felt inadequately informed by the healthcare professionals.
  Title: Lady-X Survey Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction.
  Ranges: 1-3 Best score: 1 Worst score: 3
Time Frame: At discharge
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Lady-X Survey: Information given by the healthcare professionals during childbirth.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 1 [1 to 1] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.42, Wilcoxon (Mann-Whitney)

33. Secondary Outcome: Patient Satisfaction (Lady-X Survey, Question 3)
Description: Assessed through a validated survey, Lady-X Survey. Adapted from Gartner FR, de Bekker-Grob EW et al. Calculating preference weights for the labor and delivery index: A discrete choice experiment on women's birth experiences. Value Health. 2015 Sep; 856-864.
  Question 3: Taking your wishes seriously during childbirth. Scale 1-3. 1 = Very seriously, 2 = sufficiently, 3 = insufficiently
  Title: Lady-X Survey Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction.
  Ranges: 1-3 Best score: 1 Worst score: 3
Time Frame: At discharge
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Lady-X Survey: Taking your wishes seriously during childbirth.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 1 [1 to 1] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.96, Wilcoxon (Mann-Whitney)

34. Secondary Outcome: Patient Satisfaction (Lady-X Survey, Question 4)
Description: Assessed through a validated survey, Lady-X Survey. Adapted from Gartner FR, de Bekker-Grob EW et al. Calculating preference weights for the labor and delivery index: A discrete choice experiment on women's birth experiences. Value Health. 2015 Sep; 856-864.
  Question 4: Emotional support by healthcare professionals during childbirth. Scale 1-3. 1 = Very well supported, 2 = adequately supported, 3 = inadequately supported.
  Title: Lady-X Survey Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction.
  Ranges: 1-3 Best score: 1 Worst score: 3
Time Frame: At discharge
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Lady-X Survey: Emotional support by healthcare professionals during childbirth.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 1 [1 to 1] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.75, Wilcoxon (Mann-Whitney)

35. Secondary Outcome: Patient Satisfaction (Lady-X Survey, Question 5)
Description: Assessed through a validated survey, Lady-X. Adapted from Gartner FR, de Bekker-Grob EW et al. Calculating preference weights for the labor and delivery index: A discrete choice experiment on women's birth experiences. Value Health. 2015 Sep; 856-864.
  Question 5: Feeling of security during childbirth: Scale 1-3. 1 = very safe, 2 = sufficiently safe, 3 = insufficiently safe.
  Title: Lady-X Survey Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction.
  Ranges: 1-3 Best score: 1 Worst score: 3
Time Frame: At discharge
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Lady-X Survey: Feeling of security during childbirth.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 1 [1 to 1] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney)

36. Secondary Outcome: Patient Satisfaction (Lady-X Survey, Question 6)
Description: Assessed through a validated survey, Lady-X. Adapted from Gartner FR, de Bekker-Grob EW et al. Calculating preference weights for the labor and delivery index: A discrete choice experiment on women's birth experiences. Value Health. 2015 Sep; 856-864.
  Question 6: Worries about the health of your child during childbirth. Scale 1-3; 1 = not worried, 2 = somewhat worried, 3 = very worried.
  Title: Lady-X Survey Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction.
  Ranges: 1-3 Best score: 1 Worst score: 3
Time Frame: At discharge
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Lady-X: Worries about the health of your child during childbirth.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 1 [1 to 2] | 1 [1 to 2]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney)

37. Secondary Outcome: Patient Satisfaction (Lady-X, Question 7)
Description: Assessed through a validated survey, Lady-X. Adapted from Gartner FR, de Bekker-Grob EW et al. Calculating preference weights for the labor and delivery index: A discrete choice experiment on women's birth experiences. Value Health. 2015 Sep; 856-864.
  Question 7: Time until first contact with your child. Scale 1-3. 1 = Did not take long, 2 = Took quite a long time, 3 = Took a very long time.
  Title: Lady-X Survey Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction.
  Ranges: 1-3 Best score: 1 Worst score: 3
Time Frame: At discharge
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Lady-X: Time until the first contact with your child.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 1 [1 to 1] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.24, Wilcoxon (Mann-Whitney)

38. Secondary Outcome: Patient Satisfaction (Labor Pain Scale, Question 1)
Description: Assessed through a survey (Labor pain scale). Survey assesses worst amount of pain during labor, overall amount of pain, pain associated with placement of Foley balloon, and likeliness of recommending method of induction to a friend.
  Questions 1: Worst amount of pain experienced during labor. Scale 0-100. 1 = no pain, 100 = pain as bad as it could possibly be.
  Title: Likert scale for patient satisfaction. Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction using a Likert scale. This is a way to assess from 0 to 100 patient satisfaction.
  Ranges: 0-100 Best score: 100 Worst score: 0
Time Frame: At discharge
Population: Title: Likert scale for patient satisfaction. Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction using a Likert scale. This is a way to assess from 0 to 100 patient satisfaction.
  Ranges: 0-100 Best score: 100
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Labor pain scale: Worst amount of pain that you experienced during labor.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 59.5 [40 to 85] | 70 [50 to 90]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

39. Secondary Outcome: Patient Satisfaction (Labor Pain Scale, Question 2)
Description: Assessed through a survey (Labor pain scale). Survey assesses worst amount of pain during labor, overall amount of pain, pain associated with placement of Foley balloon, and likeliness of recommending method of induction to a friend.
  Questions 2: Overall pain experienced during labor. Scale 0-100. 1 = no pain, 100 = pain as bad as it could possibly be.
  Title: Likert scale for patient satisfaction. Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction using a Likert scale. This is a way to assess from 0 to 100 patient satisfaction.
  Ranges: 0-100 Best score: 100 Worst score: 0
Time Frame: At discharge
Population: Title: Likert scale for patient satisfaction. Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction using a Likert scale. This is a way to assess from 0 to 100 patient satisfaction.
  Ranges: 0-100 Best score: 100 Worst score: 0
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Labor pain scale: Overall pain that you experienced during labor.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 50 [40 to 80.5] | 70 [50 to 87]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney)

40. Secondary Outcome: Patient Satisfaction (Labor Pain Scale, Question 3)
Description: Assessed through a survey (Labor pain scale). Survey assesses worst amount of pain during labor, overall amount of pain, pain associated with placement of Foley balloon, and likeliness of recommending method of induction to a friend.
  Questions 3: Worse amount of pain experienced during the placement of the Foley balloon. Scale 0-100. 1 = no pain, 100 = pain as bad as it could possibly be.
  Title: Likert scale for patient satisfaction. Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction using a Likert scale. This is a way to assess from 0 to 100 patient satisfaction.
  Ranges: 0-100 Best score: 100 Worst score: 0
Time Frame: At discharge
Population: as for outcome 39
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Labor pain scale: Worst amount of pain you experienced during placement of the Foley balloon.
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 20 [5 to 50] | 15 [5 to 50]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney)

41. Secondary Outcome: Patient Satisfaction (Labor Pain Scale, Question 4)
Description: Assessed through a survey (Labor pain scale). Survey assesses worst amount of pain during labor, overall amount of pain, pain associated with placement of Foley balloon, and likeliness of recommending method of induction to a friend.
  Questions 4: How likely are you to recommend your method of induction to a friend or family member. Scale 0-100. 0= very unlikely, 100= very likely.
  Title: Likert scale for patient satisfaction. Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction using a Likert scale. This is a way to assess from 0 to 100 patient satisfaction.
  Ranges: 0-100 Best score: 100 Worst score: 0
Time Frame: At discharge
Population: as for outcome 39
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Inpatient Group; Outpatient Group: Labor pain scale: How likely are you to recommend your method of induction to a friend or family member?
Arm/Group | Inpatient Group | Outpatient Group
Number analyzed (Participants) | 64 | 65
units on a scale | 99 [65 to 100] | 99 [80 to 100]
Statistical Analysis 1: Comparison: Inpatient Group vs Outpatient Group; Test type: Superiority; p = 0.60, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Enrollment to 30 days discharge
Groups:
- Inpatient Group; Outpatient Group: Adverse Events: none
Arm/Group | Inpatient Group | Outpatient Group
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/65
Serious Adverse Events (participants affected / at risk) | 16/64 | 12/65
Other Adverse Events (participants affected / at risk) | 0/64 | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inpatient Group (N=64) | Outpatient Group (N=65)
Endometritis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — Diagnosed with endometritis from admission until 30 days after discharge
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3)
Readmission within 30 days of discharge (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Umbilical cord arterial pH less than 7.1 (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1)
Umbilical cord arterial base deficit greater than 12 (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Birth injuries (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) — Birth injuries defined as cephalohematoma, subgaleal hematoma, brachial plexus injury, clavicle or humerus fracture, and scalp laceration.
Admission to the NICU (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 5 (5)

LIMITATIONS AND CAVEATS:
Results may not be generalizable to all women, safety cannot be inferred as the incidence of adverse outcomes was low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT02756689/Prot_SAP_000.pdf